CLINICAL TRIAL: NCT02121119
Title: Sciatic Popliteal Nerve Block in Foot Surgery: Lidocaine Versus Bupivacaine in Ambulatory Continuous Block With Elastomeric Pump
Brief Title: Lidocaine Versus Bupivacaine in Ambulatory Continuous Block With Elastomeric Pump
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-289
Record Dates: First submitted 2013-11-11; First posted 2014-04-23 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-09

CONDITIONS: Hallux Valgus
Keywords: Peripheral nerve block; Lidocaine; Bupivacaine
MeSH Terms: conditions — Hallux Valgus | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): 0.5% lidocaine infusion hour to 5 ml Baxter Infusor elastomeric pump 5 ml / hr.
  Interventions: Drug: Lidocaine
- Bupivacaine (Placebo Comparator): Infusion of 0.1% bupivacaine hour to 5 ml Baxter Infusor elastomeric pump 5 ml / hr.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Lidocaine — Continuous block with lidocaine in both legs. Lidocaine infusion starts 0.5% to 5 ml hour Baxter Infusor elastomeric pump LV 5 ml / hr
  Arms: Lidocaine
Drug: Bupivacaine — Continuous block with lidocaine in both legs. Infusion starts bupivacaine 0.1% to 5 ml hour Baxter Infusor elastomeric pump LV 5 ml / hr
  Other Names: Marcaine
  Arms: Bupivacaine

SUMMARY:
In practice ambulatory orthopedic surgery, one of the problems of most difficult solution is adequate control of postoperative analgesia. Pain is a frequent cause of consultation and unscheduled readmissions in this group of patients.

The use of continuous peripheral nerve blocks are an effective tool in postoperative analgesia.

In this connection, most of the studies of continuous infusions of local anesthetics by perineural catheters have been made with bupivacaine, levobupivacaine, and ropivacaine However, it has been found that lidocaine action lasts less, has lower cost and is less toxic than longer-acting agents.

The investigators aim is to compare the effectiveness of lidocaine versus bupivacaine continuous popliteal sciatic blockade ambulatory elastomeric pump.

DETAILED DESCRIPTION:
In the practice of orthopedic outpatient surgery, one of the most intractable problems is proper control of post-operative analgesia . Pain is a frequent cause of consultations and unscheduled readmissions in this group of patients.

The use of continuous peripheral nerve blocks are an effective tool in postoperative analgesia , allowing prolong the effect of the blockade by the time you want. Such techniques have been described by different groups for the management of postoperative pain with good results even successfully used in ambulatory practice .

However, sending patients home with a continuous infusion pump to local anesthetics causes some problems , such as the method of administration , cost and risk of poisoning by these drugs.

With regard to the method of administration , have been used electronic continuous infusion pumps even allow boluses of demand , with good results. However, its use implies a higher cost and are more difficult to use by patients.

An alternative of greater simplicity and lower cost is the use of disposable pumps ( elastomeric pumps ) without electronic components , which through a simple mechanism to allow a predetermined continuous infusion flow . It has been seen that the use of elastomeric pumps for continuous peripheral nerve blocks are associated with fewer technical problems and more satisfied patients electronic pumps .

Another problem that occurs with the use of ambulatory continuous technical risk is secondary to the administration of local anesthetic solutions long-acting toxicity in a home environment , without immediate medical intervention. While this is a potential risk of toxicity , this problem could be avoided by using less toxic drugs .

In this connection , most of the studies of continuous infusion of local anesthetics by perineural catheters have been made with bupivacaine , levobupivacaine , and ropivacaine . However, it has been found that lidocaine lasts less action , has a lower cost and is less toxic than the long-acting agents , although no studies which continuous infusion of lidocaine home . In addition , there is evidence of comparable effectiveness between solutions of bupivacaine and lidocaine in continuous epidural infusion for postoperative analgesia , why lidocaine is likely to be a good alternative for continuous ambulatory blocks .

Therefore, the investigators objective is to compare the effectiveness of lidocaine versus bupivacaine in ambulatory popliteal sciatic blockade with continuous elastomeric pump .

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I or II
* Body mass index between 20 and 34 kg/m2
* Bilateral surgery of ankle or foot.
* Peripheral nerve block and general anesthesia

Exclusion Criteria:

* Chronic pain.
* Illicit drug use
* Pregnancy
* Psychiatric disease
* Chronic use of analgesia
* Peripheral neuropathy
* History of severe Gastroesophageal reflux disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Resting Visual Analogue Scale average in the first 24 hours | 1 day
  Visual analogue scale

SECONDARY OUTCOMES:
Patient satisfaction | 7 days
  five point likert
Problems patient using the pump | 7 days
  Survey of local anesthetic toxicity, patient falls, catheter and exits pump problems,
Worse daily Visual Analogue Scale | 7 days
  Visual analogue scale
Number of patients using rescue analgesia and number of doses per patient | 7 days
  Milligrams of tramadol used
Resting and dynamic Visual Analogue Scale average in Post anesthesia care unit, 48, 72 hours and 7 days | 7 days
  Visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Fernando R Altermatt, MD, Principal Investigator — Assistant Professor
Locations (1):
- División de Anestesia - Facultad de Medicina Pontificia Universidad Católica, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided